CLINICAL TRIAL: NCT06270264
Title: Nociception Level Index Guidance for Analgesia in Pressure Ulcer Care in Unconscious Patients: A Pilot Study
Brief Title: Nociception Monitoring in Intensive Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111-2023
Record Dates: First submitted 2024-02-05; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Unconscious State; Pressure Ulcer
Keywords: intensive care; nociception level index; pain monitoring; pressure ulcer; palliative care
MeSH Terms: conditions — Unconsciousness; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: randomized, prospective and controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The NOL (Experimental): The caregiver nurse assessed pain by NOL monitorization along with a pain assessment tool (CPOT) and applied one mcg/kg fentanyl if NOL >25 over one minute at the monitor.
  Interventions: Device: the Nociception level index monitoring
- The Control (No Intervention): If CPOT values were still high, then one mcq/kg bolus of fentanyl at each time would be applied and repeated at five-minute intervals, if necessary, during care and 30 minutes after.

INTERVENTIONS:
Device: the Nociception level index monitoring — Nociception level index (NOL) monitoring (Medasense) is a non- invasive device differentiated from its alternatives by the use of five parameters: heart rate, heart rate variability, skin conductance level, photo-plethysmography waveform amplitude, number of skin conductance fluctuations, and their time derivatives.
  Arms: The NOL

SUMMARY:
Precisely, pain in the ICU is a multidimensional problem with a multivariate of reasons. Still, it would be simpler to manage it in unconscious palliative patients with less source of pain, but only if we can detect it practically with the help of nociception monitors. Using five parameters, nociception level index (NOL) monitoring (Medasense) is differentiated from its alternatives. Other than pain detection, this monitoring can titrate analgesic administration. This study investigates the validity of a new nociception monitoring tool, the nociception level index, and its practical impact on providing adequate analgesia in palliative patients in intensive care.

DETAILED DESCRIPTION:
The study design is randomized, prospective, and controlled in the setting of a level two intensive care unit. 40 patients (n=20) were randomized into control and nociception level. During daily pressure ulcer care, the nociception group received analgesia according to nociception level index monitorization, and the control group had the same protocol as fentanyl bolus doses of 1mcq/kg due to critical care observation pain tool assessment scores. Secondarily, hemodynamic values and variability were evaluated.

Randomization was designed by a computer-based algorithm in a 1:1 ratio into 2 (n= 20) named Group NOL and Group Control and sealed into opaque envelopes. When the inclusion/exclusion criteria are met, at the scheduled time of wound care, the caregiver nurse in the ICU chooses one envelope to apply the designed protocol for each group.

Study Intervention Caregiver nurses in the ICU were educated by the responsible doctor (B.C.) regarding the procedures after selecting study groups. In our ICU unit, routine patient care and simultaneous pressure ulcer interventions are done twice daily as day and night sessions. In our study, the caregiver nurse observed hemodynamic variables and CPOT values for pain evaluation 30 minutes before the day session of care and administered tramadol 1 mg/kg routinely. If CPOT values were still high, then one mcq/kg bolus of fentanyl at each time would be applied and repeated at five-minute intervals, if necessary, during care and 30 minutes after. Hemodynamic variables and CPOT values were noted as before, during, and after care for all patients within two groups, along with stages of pressure ulcers, and all patients had standardized care procedures. Notably, in Group NOL patients, the caregiver nurse assessed pain by NOL monitorization along with CPOT and hemodynamic variables and applied the same analgesia protocol by deciding analgesic need if NOL >25 over one minute at the monitor.

Primary outcome The total amount of analgesia for every patient was noted as the total amount of analgesic drugs used to be stated separately as tramadol and fentanyl within the period starting from 30 minutes before until 30 minutes aftercare. Although the total amount of tramadol used was in standardized protocols as 1 mg /kg, it was also investigated to refrain misevaluation due to overtreatment.

Secondary outcome Heart rate and blood pressure changes before and after care were evaluated within groups, and delta values calculated as the difference between the values at the beginning of ulcer care and before were also noted to question the effect of NOL monitorization on hemodynamic stability.

ELIGIBILITY:
Inclusion Criteria:

* Patients within the study should be followed up in the adult ICU for palliative needs of care for more than 24 hours, needing respiratory support with tracheostomy or orotracheal intubation and having pressure ulcers (less severe than stage four full-thickness pressure ulcers).

Exclusion Criteria:

* refusal to participate in the study; heart failure, atrial fibrillation and ventricular or atrial tachycardia at a level that impairs hemodynamics; continuous drug infusion for sedation and analgesia; patients with impaired peripheral perfusion and capillary refill exceeding four seconds and patients whose hemodynamics are supported by drugs such as vasopressors and inotropes.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
total fentanyl consumption | one day
  total amount of fentanyl used during pressure ulcer care session

SECONDARY OUTCOMES:
systolic blood pressure | one day
  systolic blood pressure values before, within and after care
heart rate | one day
  heart rate values before, within and after care

CONTACTS AND LOCATIONS:
Overall Officials: Berna Caliskan, MD, Principal Investigator — Anesthesiology and Reanimation Department
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gelinas C, Shahiri T S, Richard-Lalonde M, Laporta D, Morin JF, Boitor M, Ferland CE, Bourgault P, Richebe P. Exploration of a Multi-Parameter Technology for Pain Assessment in Postoperative Patients After Cardiac Surgery in the Intensive Care Unit: The Nociception Level Index (NOL)TM. J Pain Res. 2021 Dec 7;14:3723-3731. doi: 10.2147/JPR.S332845. eCollection 2021. PMID 34908872
- [Background] Shahiri TS, Richard-Lalonde M, Richebe P, Gelinas C. Exploration of the Nociception Level (NOL) Index for Pain Assessment during Endotracheal Suctioning in Mechanically Ventilated Patients in the Intensive Care Unit: An Observational and Feasibility Study. Pain Manag Nurs. 2020 Oct;21(5):428-434. doi: 10.1016/j.pmn.2020.02.067. Epub 2020 Apr 27. PMID 32354616